CLINICAL TRIAL: NCT06105762
Title: KETO-MOOD: Ketogenic Diet for Microbiome Optimization and Overcoming Depression
Brief Title: Ketogenic Diet for Depression
Acronym: KETO-MOOD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Psychiatric Clinics Basel (Network)
Responsible Party: Principal Investigator, Timur Liwinski, Doctor, University Psychiatric Clinics Basel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KET6O1L
Record Dates: First submitted 2023-10-23; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Depressive Disorder; Major Depressive Disorder; Depression, Bipolar
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Major; Bipolar Disorder | interventions — Diet, Ketogenic; Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketogenic Diet Arm (Experimental): During an 8-week period, individuals enrolled in the experimental group will undergo a low-carbohydrate, high-fat ketogenic diet intervention. We will implement the Modified Atkins Diet (MAD), which is a nutritionally rich and diverse variant of the ketogenic diet. It restricts net carbohydrate intake to less than 20g per day.
  Interventions: Other: Ketogenic Diet
- Conventional Healthy Mixed Diet Arm (Active Comparator): The control group will be provided with a standard balanced mixed diet following the recommendations for healthy nutrition by the Schweizerische Gesellschaft für Ernährung (Société Suisse de Nutrition). This diet will consist of an average daily caloric supply from carbohydrates of approximately 45 - 60%, as per the guidelines.
  Interventions: Other: Ketogenic Diet

INTERVENTIONS:
Other: Ketogenic Diet — The ketogenic diet intervention, administered as a Modified Atkins Diet, involves a significantly reduced daily carbohydrate intake, typically less than 20 grams of net carbs. This approach primarily relies on higher fat consumption to induce ketosis, a metabolic state characterized by elevated ketone body production, serving as an alternative brain fuel source.
  Other Names: LCHF (Low-Carb, High-Fat) Diet; Keto Diet; Modified Atkins Diet; Carb-Restricted Diet

SUMMARY:
Globally, it's estimated that around 300 million people are affected by depressive illness, and even with access to modern mental health care, long-term recovery is uncommon. Recently, there has been increasing interest in a promising intervention: the ketogenic diet. This diet restricts carbohydrate intake, promoting the breakdown of fats into circulating ketone bodies, which can act as an additional energy source for the brain, potentially reducing its reliance on glucose. While various sources of evidence suggest the potential benefits of the ketogenic diet for individuals with depression, robust clinical studies on its efficacy in depressed patients are lacking. Our goal is to conduct an eight-week, assessor-blinded, randomized controlled trial to investigate the therapeutic effects of a very low-carbohydrate, high-fat ketogenic diet compared to an active comparator diet in individuals with depression.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is the second leading contributor to the global burden of chronic diseases, as measured by years lived with disability. Additionally, MDD is associated with an increased risk of developing various conditions such as diabetes mellitus, heart disease, cancer, and stroke, which further adds to the disease burden. Notably, MDD significantly increases the risk of suicide, with up to 50% of the 800,000 worldwide suicides occurring during a depressive episode. The prevalence of mental disorders has been on the rise in Western societies, coinciding with the nutritional decline in typical Western diets. Traditional, nutrient-rich foods have been progressively replaced by ultra-processed foods, which are linked to heightened health risks, including type-2 diabetes, cardiovascular diseases, cancer, and depression. The ketogenic diet is a unique dietary approach that drastically limits carbohydrate intake, inducing a state of ketosis characterized by elevated levels of circulating ketone bodies. Ketone bodies, namely acetoacetate, β-hydroxybutyric acid, and acetone, are primarily produced through ketogenesis in the liver's mitochondrial matrix. Ketosis can be achieved through fasting or by consuming a low-carbohydrate diet, typically containing fewer than 20 grams of net carbs per day. Ketosis has historical roots and was a common physiological state during human evolution, particularly in the Paleolithic era when social structures were based on small groups of hunter-gatherers. In modern medicine, the ketogenic diet has been employed for nearly a century to treat refractory epilepsy. Although there is compelling evidence of the positive effects of the ketogenic diet on the brain and mental well-being, research on its effectiveness in psychiatric illnesses is still emerging. Ketosis may address various pathologies associated with depression, including frontal glucose hypometabolism, imbalances in GABA/glutamate neurotransmitter signaling, oxidative stress, mitochondrial dysfunction, inflammation (both cerebral microglial dysfunction and low-grade systemic inflammation), and perturbations in the gut microbiome. The primary hypothesis of our study is that adherence to a high-fat (≥60%) ketogenic diet, in addition to standard psychiatric care, will lead to a reduction in depressive symptoms at 4 and 8 weeks following the intervention, compared to standard psychiatric care involving a balanced mixed diet consisting of around 60% carbohydrates, with moderate amounts of fats and protein.

This study is a prospective, assessor-blinded, controlled trial with a randomized, parallel-arm design, categorized as a phase 2 trial. The focus of the study centers on a nutritional intervention as the independent variable, and it will be conducted at the University Psychiatric Clinics (UPK) in Basel, Switzerland. Participants will undergo supervised dietary training and counseling over the course of 8 weeks. The 8-week observation period is crucial for determining the effectiveness of prescribed depression treatments. Individuals eligible for the study are those who meet the diagnostic criteria for (unipolar) major depressive disorder or are currently experiencing a depressive episode within the context of bipolar affective disorder, according to ICD-10 criteria. Participants will be randomly assigned to receive either a low-carbohydrate (<20g/day) ketogenic diet or a standard balanced mixed diet. Any discussion regarding diets between assessors and patients (or trial partners) will be strictly prohibited during the trial. Dietary support will be provided, primarily in the initial days, to ensure diet adherence, address issues, and monitor potential adverse effects. Dietitians will offer guidance on setting up and maintaining the diet, utilizing recipe cards, meal planning, dietary resources, and assisting with common challenges. The MAD ketogenic diet approach will be utilized in this study, as it has shown improved adherence compared to the classic ketogenic diet, with similar anti-seizure efficacy.

The ketogenic diet presents several benefits due to its non-pharmacological nature, demonstrating safety and over a century of efficacy in epilepsy management. Emerging evidence suggests its potential advantages in addressing metabolic and neuropsychiatric conditions, potentially exceeding the effectiveness of traditional antidepressant treatments, without the associated risks of third-line interventions such as ketamine application and electroconvulsive therapy. Moreover, the ketogenic diet is cost-effective and can be self-administered by patients, enhancing their sense of self-efficacy.

ELIGIBILITY:
Inclusion criteria:

* Unequivocal diagnosis of major depressive disorder or bipolar depression according to ICD-10 and ICD-11 (as soon as approved in Switzerland) criteria
* Age ≥18 years
* The patient can give informed consent as documented by signature
* Interest in trying a dietary intervention
* Participants must refrain from using any non-prescribed psychotropic agents during the study period including alcohol and illicit drugs such as cannabis; long term pain medication, caffeine and nicotine are excluded from that rule

Exclusion criteria:

* Inability to follow the study procedures, e.g., because of a language barrier, neurological and interfering mental disorders, dementia
* Anorexia nervosa
* BMI <18.5 kg/m2
* Pregnancy or breast feeding
* Current electroconvulsive therapy (ECT)
* Concurrent ketamine therapy
* Inability to follow the procedures of the study, e.g. due to language barrier, neurological and interfering mental disorders, high-grade dementia, etc.
* Porphyria
* Type 1 diabetes
* Insulin-dependent type 2 diabetes
* Contraindicated medical conditions; besides rare hereditary metabolic disorders (typically diagnosed in childhood), contraindications comprise acute pancreatitis, nephrolithiasis, advanced renal failure, advanced liver failure, advanced congestive heart failure, advanced pulmonary disease with respiratory failure, and concurrent use of SGLT2 inhibitors

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Depressive Symptoms Severity | Baseline (week 0), week 4, week 8
  * Assessment Tool: Hamilton Depression Rating Scale (HAM-D17)
  * Scale Range: 0 to 54 (higher scores indicate more severe depressive symptoms)

SECONDARY OUTCOMES:
Anxiety Symptoms Severity | Baseline (week 0), week 4, week 8
  * Assessment Tool: Generalized Anxiety Disorder-7 (GAD-7)
  * Scale Range: 0-21 (higher scores indicate greater severity of anxiety symptoms)
Functioning | Baseline (week 0), week 4, week 8
  * Assessment Tool: Clinical Global Impression (CGI)
  * Scale Range: 1-7 (higher scores indicate poorer functioning)
Hedonic Tone | Baseline (week 0), week 4, week 8
  - Assessment Tool: Snaith-Hamilton Pleasure Scale (SHAPS)
Sleep Quality | Baseline (week 0), week 4, week 8
  - Assessment Tool: Insomnia Severity Index (ISI)
Subjective Depressive Symptom Burden | Baseline (week 0), week 4, week 8
  - Assessment Tool: Beck Depression Inventory II
Changes in Serum Levels of Brain-Derived Neurotrophic Factor (BDNF) | Baseline (week 0), week 4, week 8
  * Assessment Tool: Enzyme-Linked Immunosorbent Assay (ELISA)
  * Measuring BDNF levels in plasma using ELISA
Changes in Serum Level of Highly Sensitive C-Reactive Protein (hsCRP) | Baseline (week 0), week 4, week 8
  - Assessment Tool: Ultrasensitive ELISA
Changes in Fecal Metagenomics Shotgun Sequencing | Baseline (week 0), week 8
  * Assessment Tool: Fecal metagenomics shotgun sequencing
  * Analyzing fecal samples via shotgun sequencing to determine gut microbiota composition and diversity
Changes in Serum Metabolomics Profile | Baseline (week 0), week 8
  - Assessment Tool: Liquid Chromatography-Mass Spectrometry (LC-MS)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Francis H, Stevenson R. The longer-term impacts of Western diet on human cognition and the brain. Appetite. 2013 Apr;63:119-28. doi: 10.1016/j.appet.2012.12.018. Epub 2013 Jan 3. PMID 23291218
- [Result] Gangwisch JE, Hale L, Garcia L, Malaspina D, Opler MG, Payne ME, Rossom RC, Lane D. High glycemic index diet as a risk factor for depression: analyses from the Women's Health Initiative. Am J Clin Nutr. 2015 Aug;102(2):454-63. doi: 10.3945/ajcn.114.103846. Epub 2015 Jun 24. PMID 26109579
- [Result] Wheless JW. History of the ketogenic diet. Epilepsia. 2008 Nov;49 Suppl 8:3-5. doi: 10.1111/j.1528-1167.2008.01821.x. PMID 19049574
- [Result] Mentzelou M, Dakanalis A, Vasios GK, Gialeli M, Papadopoulou SK, Giaginis C. The Relationship of Ketogenic Diet with Neurodegenerative and Psychiatric Diseases: A Scoping Review from Basic Research to Clinical Practice. Nutrients. 2023 May 11;15(10):2270. doi: 10.3390/nu15102270. PMID 37242153
- [Result] Smolensky IV, Zajac-Bakri K, Gass P, Inta D. Ketogenic diet for mood disorders from animal models to clinical application. J Neural Transm (Vienna). 2023 Sep;130(9):1195-1205. doi: 10.1007/s00702-023-02620-x. Epub 2023 Mar 21. PMID 36943505
- [Result] Norwitz NG, Sethi S, Palmer CM. Ketogenic diet as a metabolic treatment for mental illness. Curr Opin Endocrinol Diabetes Obes. 2020 Oct;27(5):269-274. doi: 10.1097/MED.0000000000000564. PMID 32773571